CLINICAL TRIAL: NCT01885416
Title: The Impact of Dairy Products on Postprandial Inflammation in Obese Males
Brief Title: Impact of Dairy Products on Postprandial Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agroscope Liebefeld-Posieux Research Station ALP (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Guy Vergeres, Dr., Agroscope Liebefeld-Posieux Research Station ALP
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUTRICHIP-2
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Inflammation; Obesity; Nutritional Intervention
MeSH Terms: conditions — Inflammation; Obesity | interventions — Dairy Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high fat meal without dairy products (Active Comparator): high fat meal without dairy products
  Interventions: Other: consumption of high fat test meal without dairy products
- high fat meal with additional milk (Experimental): high fat meal with additional milk
  Interventions: Other: consumption of high fat test meal with dairy products
- dairy product meal (Experimental): dairy product meal
  Interventions: Other: consumption of test meal based on dairy products

INTERVENTIONS:
Other: consumption of test meal based on dairy products
  Arms: dairy product meal
Other: consumption of high fat test meal without dairy products
  Arms: high fat meal without dairy products
Other: consumption of high fat test meal with dairy products
  Arms: high fat meal with additional milk

SUMMARY:
The study will quantitatively evaluate the systemic, postprandial inflammatory and metabolic response to the ingestion of three different meals in obese subjects. The administered meals will differ in the proportion of dairy products. Postprandial response will be monitored during 6 hours after meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* male
* BMI ≥ 20 kg/m2
* age 25-55 y
* informed consent

Exclusion Criteria:

* Physiological or psychological diseases
* Allergies to food or intolerance to high-fat meal
* Vegetarians
* Chronic intake of drugs
* Smokers
* Diabetes mellitus Type I and II
* Debilitating kidney diseases
* Debilitating liver diseases
* Clinically established coronary heart diseases
* Ingestion of vitamins or dietary supplements during the course of the study

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Inflammation markers in blood plasma (IL-6, TNF-alpha) | 0,6h

SECONDARY OUTCOMES:
Biomarkers in blood (serum insulin, plasma glucose, GLP-1, lipids) | 0,1,2,4,6h
Endotoxin in blood serum | 0,6h

OTHER OUTCOMES:
Blood cell transcriptome | 0,2,4,6h
blood serum metabolome | 0,2,4,6h

CONTACTS AND LOCATIONS:
Overall Officials: Kur Laederach, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Alexandra Schmid, Study Director — Agroscope Liebefeld-Posieux ALP; Caroline Buri, MD, PhD, Study Director — Insel Gruppe AG, University Hospital Bern; Guy Vergères, PhD, Study Director — Agroscope Liebefeld-Posieux ALP
Locations (1):
- University Hospital, Inselspital Berne, Bern, Canton of Bern, Switzerland